CLINICAL TRIAL: NCT06475313
Title: Risk Assessment of Proximal Contact Loss Between Implant-supported Prostheses and Adjacent Teeth.
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20240613-05
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
Keywords: food impaction; proximal contact loss; Implant supported prosthesis; Dentition defect; risk factors
MeSH Terms: conditions — Peri-Implantitis | interventions — short-wavelength opsin; Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: plaque index assessment, periodontal probing, Bleeding on probing (BOP), Prosthetic adjacency check, initial occlusal contact, maximum occlusal contact, and filling of the cusps. — oral panoramic radiograph
  Other Names: Radiation

SUMMARY:
In this study, we collected and analysed the review results of 100 patients over 18 years of age who received implant fixed restorations in the Department of Stomatology of the First Hospital of Nanjing, China. The aim was to investigate the incidence of loss of contact between implant restorations and adjacent teeth and its influencing factors. Our findings may provide better insights for treatment planning and prevention of PCL.

DETAILED DESCRIPTION:
Food impaction is a common complication after implant-supported restorations. Several studies have reported that more than 40%-66.9% of patients feel food impaction between the implant restoration and adjacent natural teeth. The most common cause of food impaction after implant restoration is the proximal contact loss(PCL), which has been reported to occur in 34% to 65% of cases. The location of PCL creates discomfort and leads to gingival inflammation and even peri-implant bone resorption, which ultimately leads to loosening of the implant. In our long-term clinical observation, not all final restorations suffer from PCL. The occurrence of PCL may be related to a number of factors such as age, gender, functional time, and so on. However, the literature addressing this issue is still limited. In this study, we collected and analysed the review results of selected patients who underwent implant-supported restorations in the First Hospital of Nanjing, China, to investigate the incidence of PCL between the implant restorations and the adjacent teeth adjacent , and the factors influencing it. Our findings may provide better insights for treatment planning and prevention of PCL.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients over the age of 18, can fully understand the nature of the proposed and be able to sign a consent form.
* (2) patients who underwent dental implant surgery and delivered prostheses for more than 3 months in Nanjing First Hospital.

Exclusion Criteria:

* (1) The implant site or adjacent teeth were severely injured and the adjacent teeth were extracted;
* (2) the same quadrant orthodontic or splint treatment;
* (3) the prostheses have been removed due to failure or need further treatment;
* (4) implant-supported prostheses in both mesial and distal sites;
* (5) the adjacent teeth were directly or indirectly fixed with the implant-supported prosthesis;
* (6) patients with missing clinical records of PD, PCR and BOP.
* (7) The prosthetic prosthesis with implant-supported prosthesis was delivered for less than 3 months in Nanjing First Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: One hundred consecutive patients, who had received either implant-supported fixed partial denture (FPD) or implant-supported single crown (SC) in the posterior region and were under regular review, were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
the proximal contact surface was adjusted by a dental floss (Reach waxed dental floss from Johnson & Johnson, standard thickness) | Patients with implant-supported prostheses reviewed 3 months after delivery were eligible for inclusion in this study.
  The degree of proximal contact loss(PCL) was evaluated with a dental floss passing through the contact areas and classified as: (a) tight: sufficient resistance to the passage of the floss; (b) loose: insufficient resistance to the passage of the floss; and (c) open: contact: no resistance to the passage of the floss. The presence of an open or loose contact was classified as PCL.

SECONDARY OUTCOMES:
oral panoramic radiograph | Patients with implant-supported prostheses reviewed 3 months after delivery were eligible for inclusion in this study.
  Using the radiograph analysis software's measuring function, the amount of alveolar bone resorption of the implant as well as adjacent teeth was evaluated. (a)The original bone height was measured as the distance between the enamel-cemental junction and the root apex (or the implant neck edge and the implant base). (b)The existing bone height was measured as the distance between the top of the alveolar ridge to the root apex. (c) The height of alveolar bone resorption was calculated by subtracting the original bone height from the existing bone height.
Bausch Arti-Fol R metallic Shimstock-Film | Patients with implant-supported prostheses reviewed 3 months after delivery were eligible for inclusion in this study.
  (a) Initial occlusal contact: Bausch articulating paper was applied to the restoration's occlusal surface, the patient was told to close their mouth slowly, the teeth just gently touched, and they opened their mouth right away. The paper was then removed, and the restoration's occlusal surface was examined to see if it had left a red mark. (b) Final occlusal contact: If the patient's restoration and opposing jaw teeth do not make contact during the initial occlusion, place the Bausch articulating paper on the restoration's occlusal surface, ask them to clench their teeth, and then have them open their mouth, take the paper out, and check to see if the implant's occlusal surface has any marks on it.

CONTACTS AND LOCATIONS:
Overall Officials: Changao Xue, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Ning Luo, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Juan Lin, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Information about participants in this study will not be shared with investigators outside the study, and all study participants are identified by initials.

REFERENCES:
- [Background] Yen JY, Kang L, Chou IC, Lai YL, Lee SY. Risk assessment of interproximal contact loss between implant-supported fixed prostheses and adjacent teeth: A retrospective radiographic study. J Prosthet Dent. 2022 Jan;127(1):86-92. doi: 10.1016/j.prosdent.2020.06.023. Epub 2020 Nov 7. PMID 33172648
- [Background] Bompolaki D, Edmondson SA, Katancik JA. Interproximal contact loss between implant-supported restorations and adjacent natural teeth: A retrospective cross-sectional study of 83 restorations with an up to 10-year follow-up. J Prosthet Dent. 2022 Mar;127(3):418-424. doi: 10.1016/j.prosdent.2020.09.034. Epub 2020 Dec 17. PMID 33342612
- [Background] Liang CH, Nien CY, Chen YL, Hsu KW. The prevalence and associated factors of proximal contact loss between implant restoration and adjacent tooth after function: A retrospective study. Clin Implant Dent Relat Res. 2020 Jun;22(3):351-358. doi: 10.1111/cid.12918. Epub 2020 May 17. PMID 32419242
- [Background] Gasser TJW, Papageorgiou SN, Eliades T, Hammerle CHF, Thoma DS. Interproximal contact loss at implant sites: a retrospective clinical study with a 10-year follow-up. Clin Oral Implants Res. 2022 May;33(5):482-491. doi: 10.1111/clr.13908. Epub 2022 Mar 1. PMID 35194854